CLINICAL TRIAL: NCT05924815
Title: A Randomized, 2-Part, Single-Dose, Crossover Study to Evaluate the Effect of Aficamten Administration on QT/QTc Interval in Healthy Participants
Brief Title: Study to Evaluate the Effect of Aficamten Administration on QT/QTc Interval
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: CY 6019
Record Dates: First submitted 2023-06-07; First posted 2023-06-29 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Healthy Participants
Keywords: CK-3773274; CK-274; Aficamten
MeSH Terms: interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- Part A (Dose Finding Cohort 1): Aficamten 50 mg (Experimental): Participants in this arm will receive a single oral dose of 50 mg aficamten.
  Interventions: Drug: Aficamten
- Part A (Dose Finding Cohort 2): Aficamten 75 mg (Experimental): Participants in this arm will receive a single oral dose up to 75 mg aficamten.
  Interventions: Drug: Aficamten
- Part A (Dose Finding Cohort 3): Aficamten 100 mg (Experimental): Participants in this arm will receive a single oral dose up to 100 mg aficamten.
  Interventions: Drug: Aficamten
- Part B (TQT Study): Aficamten (Experimental): Participants will receive a single oral dose of aficamten. The dose will be determined based on review of Part A PK parameters, echocardiogram parameters, safety, and tolerability for aficamten.
  Interventions: Drug: Aficamten
- Part B (TQT Study): Aficamten-matching Placebo (Placebo Comparator): Participants in this arm will receive a single oral dose of aficamten-matching placebo.
  Interventions: Drug: Aficamten-matching Placebo
- Part B (TQT Study): Moxifloxacin 400 mg (Active Comparator): Participants will receive a single oral dose of 400 mg moxifloxacin
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: Aficamten — Oral Tablet
  Arms: Part A (Dose Finding Cohort 1): Aficamten 50 mg; Part A (Dose Finding Cohort 2): Aficamten 75 mg; Part A (Dose Finding Cohort 3): Aficamten 100 mg; Part B (TQT Study): Aficamten
Drug: Aficamten-matching Placebo — Oral Tablet
  Arms: Part B (TQT Study): Aficamten-matching Placebo
Drug: Moxifloxacin — Oral Tablet
  Arms: Part B (TQT Study): Moxifloxacin 400 mg

SUMMARY:
This is a single-center, 2-part (Part A and Part B) study in healthy participants. Part A (Dose Finding) is an open-label, SAD study to identify the dose for Part B. Part B (TQT Study) is a randomized, double-blind (with respect to aficamten and matching placebo), positive- and placebo-controlled, single-dose, 3-way crossover study to evaluate the effect of aficamten administration on QT/QTc interval.

ELIGIBILITY:
Inclusion Criteria:

* Healthy, adult, male or female, 18-45 years of age, inclusive, at the screening visit.
* Continuous non-smoker who has not used nicotine- and tobacco -containing products for at least 3 months prior to the first dosing based on participant self- reporting.
* Body mass index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2 at the screening visit.
* Medically healthy with no clinically significant medical history, physical examination, laboratory profiles, and vital signs, as deemed by the PI or designee, including the following:

  * Supine blood pressure is ≥ 90/40 mmHg and ≤ 140/90 mmHg at the screening visit.
  * Oxygen saturation (SpO2) is ≥ 95% at the screening visit.
  * Liver function tests (e.g., bilirubin, aspartate aminotransferase [AST], alanine aminotransferase [ALT]) considered not clinically significant in the opinion of the PI or designee at the screening visit.
  * Estimated creatinine clearance ≥ 90 mL/min at the screening visit.
* No clinically significant history and presence of ECG findings as judged by the PI or designee at the screening visit and first check-in, including each of the following:

  * HR between 50 bpm and 100 bpm, inclusive.
  * QTcF interval is ≤450 msec (males) and ≤460 msec (females).
  * QRS ≤110 msec; if >110 msec, result will be confirmed by a manual over read.
  * PR ≤220 msec.
* LVEF ≥65% at the screening visit.

Exclusion Criteria:

* History of any illness that, in the opinion of the PI or designee, might confound the results of the study or poses an additional risk to the participant by their participation in the study.
* History or presence of alcohol or drug abuse within the past 2 years prior to the first dosing.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2023-05-15 (Actual); Primary Completion 2023-11-14 (Actual); Study Completion 2023-11-14 (Actual)

PRIMARY OUTCOMES:
Part A: To determine the dose for Part B | Baseline to End of Study, up to 8 weeks
  To determine the dose for Part B based on Part A PK and safety data.
Part B: placebo-corrected dQTcF for aficamten | Baseline to End of Study, up to 14.5 weeks
  To evaluate the effect of a single oral dose of aficamten on the QTc interval in healthy participants.

SECONDARY OUTCOMES:
Part B: placebo-corrected dQTcF for moxifloxacin | Baseline to End of Study, up to 14.5 weeks
  To demonstrate assay sensitivity of the study to detect a small QTc effect using moxifloxacin as a positive control in healthy participants.

CONTACTS AND LOCATIONS:
Overall Officials: Cytokinetics, MD, Study Director — Cytokinetics
Locations (1):
- Celerion, Inc 2420, Tempe, Arizona, United States

IPD SHARING:
Plan to Share IPD: No